CLINICAL TRIAL: NCT00731653
Title: An Open-Label Extension Study to Assess the Tolerability of BCI-024 in Combination With BCI-049 in Patients With Major Depressive Disorder
Brief Title: Open Label Extension Assessing the Tolerability of BCI-024 in Combination With BCI-049 in Patients With Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: BrainCells Inc. (Industry)
Responsible Party: Principal Investigator, Maurizio Fava, MD, Fava, Maurizio, MD, Massachusetts General Hospital
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBM-IT-01-EXT
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Results first posted 2013-12-17 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-10

CONDITIONS: Major Depressive Disorder
Keywords: depression; combination
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): BCI-024 and BCI-049
  Interventions: Drug: Combination Product: BCI-024 + BCI-049

INTERVENTIONS:
Drug: Combination Product: BCI-024 + BCI-049 — BCI-024 and BCI-049 once a day at bedtime for 6 weeks

SUMMARY:
The objective of this study is to allow patients who have participated in the precursor study of BCI-024 in combination with BCI-049 versus placebo or BCI-024 alone (Protocol #CBM-IT-01) to receive 6 weeks of open-label treatment with an increased dose of BCI-024 in combination with an increased dose of BCI-049.

The safety and tolerability of this higher dose of the combination will be evaluated, as will the treatment effect in reducing symptoms of depression in patients with MDD.

DETAILED DESCRIPTION:
Up to approximately 120 adult outpatients meeting the study's inclusion and exclusion criteria may be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are willing to provide written informed consent and who have completed participation in Protocol CBM-IT-01 are eligible for the study.
* Eligible subjects will have demonstrated compliance with all CBM-IT-01's protocol requirements.

Exclusion Criteria:

- Subjects who did not complete their participation in Protocol CBM-IT-01 are not eligible for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2008-07; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Fava, MD, Principal Investigator — Massachusetts General Hospital; Andrew A Nierenberg, MD, Principal Investigator — Massachusetts General Hospital
Locations (9):
- United States (9):
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - Synergy Research Centers, San Diego, California
  - Atlanta Institute of Medicine & Research, Inc., Altanta, Georgia
  - Capital Clinical Research Associates, Rockville, Maryland
  - NorthCoast Clinical Trials, Beachwood, Ohio
  - CRI Worldwide, Philadelphia, Pennsylvania
  - FutureSearch Clinical Trials, L.P., Austin, Texas
  - FutureSearch Trials of Dallas, L.P., Dallas, Texas
  - Claghorn-Lesem Research Clinic, Ltd., Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Following their participation in the CBM-IT-01 study, subjects were offered the opportunity to participate in this open-label extension study. The study was conducted 9 study centers between June 2008 and February 2009.
Groups:
- BCI-024 and BCI-049 (Buspirone and Melatonin): BCI-024 (Buspirone)30 mg QD and BCI-049 (Melatonin) 6 mg QD Open-label
Period: Overall Study
Arm/Group | BCI-024 and BCI-049 (Buspirone and Melatonin)
Started | 81
Completed | 72
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | BCI-024 and BCI-049 (Buspirone and Melatonin)
Number analyzed (Participants) | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 81
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 43.7 (11.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 81

OUTCOME MEASURES:

1. Primary Outcome: The Primary Safety and Tolerability Outcome Measure is Reported Adverse Events.
Time Frame: Weeks 0-6 (study treatment) and Weeks 7 and 8 (post-treatment)
Population: All patients who received at least one dose of study treatment during the extension phase were included in the analysis population. Analyses were performed with observed data. Tables and listings of safety and efficacy assessments will include all data observed. There was no imputation or adjustment for missing data values.
Measure: Number; unit: participants
Arm/Group | BCI-024 and BCI-049 (Buspirone and Melatonin)
Number analyzed (Participants) | 81
participants | 81

ADVERSE EVENTS:
Arm/Group | BCI-024 and BCI-049 (Buspirone and Melatonin)
Serious Adverse Events (participants affected / at risk) | 0/81
Other Adverse Events (participants affected / at risk) | 42/81
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCI-024 and BCI-049 (Buspirone and Melatonin) (N=81)
Headache (Nervous system disorders) | 13 (14)
Somnolence (Nervous system disorders) | 6 (6)
Dizziness (Nervous system disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Dry Mouth (Gastrointestinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
This was an open-label study. Conclusions regarding the efficacy of the combination study drug were not made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No